CLINICAL TRIAL: NCT01009528
Title: Development and Evaluation of Electronic Feedback, a Tool for Quality Assurance of the Diabetic Care in General Practice
Brief Title: Electronic Feedback on Diabetic Care to General Practitioners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Trine Guldberg,MD, Institute of Public Health, Aarhus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2008-41-2792
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2009-11-09 (Estimated); Status verified 2009-11

CONDITIONS: Type 2 Diabetes
Keywords: Quality of care; General Practice; Electronic Feedback System
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Admission to electronic feedback system
  Interventions: Device: Electronic feedback system on diabetes care
- control (No Intervention): Control group. No special attention

INTERVENTIONS:
Device: Electronic feedback system on diabetes care — An electronic feedback system was introduced in randomized primary care clinics providing an overview of quality of care. The intervention ran for 15 months.
  Other Names: Electronic feedback system; Decission support system
  Arms: Intervention

SUMMARY:
The aim of this study is to determine whether electronic feedback to general practitioners on quality of Type 2-Diabetes care increases the quality of care measured on process and outcome measures contained in the national guidelines. Effect evaluation will be performed using a mixed method design.

DETAILED DESCRIPTION:
Background: In an effort to optimize diabetes care in general practice, an electronical feedback system has been developed. The system will be evaluated both quantitative and qualitative.

Method: The general practitioners (GP´s) of the Region of Southern Denmark have been randomised to either admission or no admission to the electronic feedback system. The system was launched 1/3-2007 and ran for one year prior to evaluation.

Quantitative evaluation by assessment of the following end-points: Patients Hba1c-level, number of patients who have had their hba1c-level measured within the last year, cholesterol-level and number of patients who have had an eye examination within the last year.

Qualitative evaluation by interviewing GP´s who have had admission to the system.

Qualitative data have been collected through interviews with intervention GPs, designed to uncover motivational factors as well as barriers concerning the use of feedback on chronic care in general practice. Data are being analyzed.

Quantitative data are being gathered. Perspective: This project will shed light on the value of electronic feedback systems within chronic care in general practice.

Based on this project it will be possible to set up a system for automatic electronic monitoring and feedback of the quality of care in general practice, taking motivational factors of the GP s into account during implementation.

ELIGIBILITY:
Inclusion Criteria:

* Prevalent Type 2-diabetes as confirmed by Primary Care Physician.
* Patient alive throughout the intervention period.
* GP actively working throughout the intervention period (not retired).

Exclusion criteria:

* death during intervention
* moved out of geographic area during intervention
* GP retired during intervention

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2458 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Outcome and process measures from the danish diabetes guideline | 1/3 2007-1/6 2008

SECONDARY OUTCOMES:
Interview data concerning the impact of the electronic feedback system in the intervention clinics | 1/3 2007-1/6 2008

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Lauritzen, MD, Dr. Med., Study Director — Professor
Locations (1):
- Dept. of General Medicine, Institute of Public Health, Aarhus University, Aarhus, Denmark

REFERENCES:
- [Background] Guldberg TL, Lauritzen T, Kristensen JK, Vedsted P. The effect of feedback to general practitioners on quality of care for people with type 2 diabetes. A systematic review of the literature. BMC Fam Pract. 2009 May 6;10:30. doi: 10.1186/1471-2296-10-30. PMID 19419548
- [Derived] Guldberg TL, Vedsted P, Kristensen JK, Lauritzen T. Improved quality of Type 2 diabetes care following electronic feedback of treatment status to general practitioners: a cluster randomized controlled trial. Diabet Med. 2011 Mar;28(3):325-32. doi: 10.1111/j.1464-5491.2010.03178.x. PMID 21309841
- [Derived] Guldberg TL, Vedsted P, Lauritzen T, Zoffmann V. Suboptimal quality of type 2 diabetes care discovered through electronic feedback led to increased nurse-GP cooperation. A qualitative study. Prim Care Diabetes. 2010 Apr;4(1):33-9. doi: 10.1016/j.pcd.2010.01.001. Epub 2010 Jan 21. PMID 20096659